CLINICAL TRIAL: NCT04626895
Title: Measuring the Efficacy of Paxman Scalp Cooling to Prevent Chemotherapy Induced Alopecia (CIA) in Black Patients With Stage I-III Breast or Gynecological Cancers
Brief Title: Efficacy of Paxman Scalp Cooling to Prevent Chemo Induced Alopecia in Black Patients With Breast or GYN Cancers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medstar Health Research Institute (Other)
Collaborators: Paxman (Unknown)
Responsible Party: Principal Investigator, Asma Dilawari, Assistant Professor of Medicine, Medstar Health Research Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00000334
Record Dates: First submitted 2020-10-28; First posted 2020-11-13 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Breast Cancer; Ovarian Cancer; Gynecologic Neoplasm; Endometrial Cancer
MeSH Terms: conditions — Breast Neoplasms; Ovarian Neoplasms; Genital Neoplasms, Female; Endometrial Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Scalp Cooling (Other): Patients who be will using the scalp cooling device during chemotherapy will be enrolled in tis arm
  Interventions: Device: Paxman Scalp Cooling Device
- Non Scalp-Cooling (No Intervention): Patients who do not use scalp cooling device during chemotherapy will be enrolled in this arm.

INTERVENTIONS:
Device: Paxman Scalp Cooling Device — Paxman scalp cooling device
  Arms: Scalp Cooling

SUMMARY:
This study will measure the efficacy of scalp cooling with the Paxman Scalp Cooling (PSC) device in a diverse patient population with success measured as prevention of more than 50% hair loss during chemotherapy. We propose that scalp cooling has distinct efficacy in participants with black or ethnic-minority hair types due to differences in textures, hair thickness. This study will examine the success rate of scalp cooling in black patients receiving chemotherapy for breast or gynecological cancer.

DETAILED DESCRIPTION:
The primary objective is to measure the efficacy of the PSC device in preventing CIA in this diverse patient population with success measured as prevention of >grade 2 alopecia by self-report using the modified Dean scale or the VAS scale in >50% of participants using the intervention. We propose that scalp cooling has distinct efficacy in participants with black or ethnic-minority hair types due to differences in textures, hair thickness.

The study aims include delivery of scalp cooling at each chemotherapy cycle with measurements of CIA at assigned intervals using patient self-report measured by the modified Dean scale and the Visual Analog Scale (VAS) outlined below.

The secondary aims are provider assessments of alopecia as measured by the NCI grading scale of alopecia, adverse effects of scalp cooling procedures such as headaches, dizziness, and pain, reasons for refusal or drop-out of study intervention.

Psychosocial and quality-of- life (QOL) effects of CIA in study participants will be measured using patient reported outcomes. The EORTC QLQ-B45 and Chemotherapy-Induced-Alopecia-Distress Scale (CADS) will be administered at designated time intervals.

ELIGIBILITY:
Inclusion Criteria:

* Stage I-III breast cancer patients
* Stage I-III endometrial cancer patients
* Stage I-III ovarian cancer patients
* Self-identified as black: African, African-American, or Caribbean black are included . Patients of mixed race who identify as black are also included.
* Planned for >4 cycles of chemotherapy in the neoadjuvant or adjuvant setting with curative intent
* At least one chemotherapy agent being a taxane.
* Ability to read and answer questions in English
* Ability to sign informed consent for themselves.
* Able to fit into one of available cap sizes

Exclusion Criteria:

* Metastatic cancer patients
* Patients who do not self-identify as black (see definition above)
* History of cryoglobulinemia or cold agglutin disease
* Prior chemotherapy
* Non-taxane chemotherapy regimens (anthracycline based chemotherapy regimens are eligible for breast cancer patients)
* Baseline alopecia
* Concurrent medications to prevent hair loss
* Cold urticaria and cold- induced anaphylaxis
* Unable to fit into an available cap size
* Adults unable to consent on their own will not be eligible
* Individuals unable to answer questionnaires in English will not be eligible.
* Pregnant women will not be permitted to enroll as the use of this device in pregnancy is not well studied
* Prisoners will not be included in this study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-06-04 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Patient reported rate of alopecia rate of alopecia | During active chemotherapy and completion of study, an average of 6 months
  Patient-reported rate of alopecia as measured by the modified Dean Scale and VAS. Hair preservation is defined in this scale as <50% hair loss (< grade 2) or score of <50 on VAS

SECONDARY OUTCOMES:
Psychosocial assessments of chemotherapy-induced alopecia | During active chemotherapy and completion of study, an average of 6 months
  Psychosocial assessments of chemotherapy-induced alopecia will be measured by validated CADS (Chemotherapy-induced Alopecia Distress Scale) at designated time intervals. The questionnaire is composed of a 4-point likert Scale and 4 multi-items distress domain that include Physical (2 questions), Emotional (6 questions), Activity (6 questions) and Relationship (1 question). A score of 4 for each domain indicates greater distress. A score of 1 represents no distress.
Quality of life assessments of chemotherapy-induced alopecia | During active chemotherapy and completion of study, an average of 6 months
  Quality of life assessments of chemotherapy-induced alopecia will be measured by EORTC QLQ BR45 questionnaire at designated time intervals. Higher score (4 for each question) is worse.

CONTACTS AND LOCATIONS:
Overall Officials: Asma Dilawari, MD, Principal Investigator — Medstar Health Research Institute
Locations (1):
- MedStar Washington Hospital Center, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: Yes
Study protocol, statistical analysis plan, informed consent form, clinical study report and analytic code will be shared.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Now until 5 years.
Access Criteria: De-identified outcomes measures and analyses will be shared.

REFERENCES:
- [Derived] Dilawari A, Gallagher C, Alintah P, Chitalia A, Tiwari S, Paxman R, Adams-Campbell L, Dash C. Does Scalp Cooling Have the Same Efficacy in Black Patients Receiving Chemotherapy for Breast Cancer? Oncologist. 2021 Apr;26(4):292-e548. doi: 10.1002/onco.13690. Epub 2021 Feb 17. PMID 33512741